CLINICAL TRIAL: NCT05581875
Title: A Phase 1/2, Dose and Schedule Evaluation Study to Investigate the Safety and Clinical Activity of Belantamab Mafodotin Administered in Combination With Daratumumab, Pomalidomide and Dexamethasone in Patients With Relapsed/ Refractory Multiple Myeloma Previously Treated With One Line of Therapy Who Are Lenalidomide Refractory.
Brief Title: A Study to Investigate the Safety and Clinical Activity of Belantamab Mafodotin in Combination With Daratumumab, Pomalidomide and Dexamethasone in Patients With Relapsed/ Refractory Multiple Myeloma Previously Treated With One Line Therapy Who Are Lenalidomide Refractory
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hellenic Society of Hematology (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: EAE127
Record Dates: First submitted 2022-10-05; First posted 2022-10-17 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Multiple Myeloma; Multiple Myeloma in Relapse; Neoplasms; Gammopathy, Monoclonal; Paraproteinemias; Blood Protein Disorders; Haematologic Disease; Corneal Disease; Neoplasms, Plasma Cell
MeSH Terms: conditions — Multiple Myeloma; Neoplasms; Paraproteinemias; Blood Protein Disorders; Hematologic Diseases; Corneal Diseases; Neoplasms, Plasma Cell | interventions — daratumumab; pomalidomide; Dexamethasone

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part 1 : Dose finding (Experimental): Belantamab mafodotin will be administered by intravenous infusion as a combination therapy as a calculated dose on Day 1 of every other 28-day cycle.
  Belantamab mafodotin starting dose for Part 1:
  * Cohort 1: 1.4 Q8W = 1.4 mg/kg on Day 1 of every other 28-day cycle
  * Cohort 2: 1.9 Q8W = 1.9 mg/kg on Day 1 of every other 28-day cycle
  Daratumumab 1800mg SC (fixed dose) on:
  Cycles 1-2: days 1, 8, 15, 22 Cycles 3-6: days 1, 15 Cycles 7+: day 1
  Pomalidomide: 4 mg/d on days 1-21 of every 28-day cycle.
  Dexamethasone: 40 mg/d on days 1, 8, 15, 22 of every 28-day cycle in participants < 75 years; 20 mg/d on days 1, 8, 15, 22 of every 28-day cycle in participants ≥ 75 years.
  Interventions: Drug: Belantamab Mafodotin-Blmf; Drug: Daratumumab; Drug: Pomalidomide; Drug: Dexamethasone

INTERVENTIONS:
Drug: Belantamab Mafodotin-Blmf — Blmf will be available as 100 mg/vial in single-use vial for reconstitution, supplied as lyophilized powder. Blmf will be delivered as IV solution over at least 30 minutes
Drug: Daratumumab — Daratumumab will be administered with subcutaneous injections. On days where Blmf is given together with daratumumab, daratumumab should be performed first.
Drug: Pomalidomide — Pomalidomide will be administered per os.
Drug: Dexamethasone — Dexamethasone will be administered intravenously or per os.

SUMMARY:
This is a phase 1/2, open label, single-center study designed to assess the safety and preliminary clinical activity of different belantamab mafodotin doses in combination with daratumumab, pomalidomide, and dexamethasone (DPd) in patients with Relapsed/ Refractory Multiple Myeloma (RRMM) previously treated with one line of therapy who are lenalidomide refractory.

This will be a 2-Part study. Part 1 will evaluate the safety of belantamab mafodotin in combination with DPd in 2 cohorts and determine the Recommended Phase 2 Dose (RP2D). In the dose expansion phase (Part 2) an expansion cohort will be treated with the RP2D. The expansion cohort will randomize participants (1:1) in two groups to evaluate two alternate dose modification guidelines for corneal AEs. Part 2 will further evaluate the safety and assess the preliminary clinical activity of the belantamab mafodotin RP2D in combination with DPd.

Overall, approximately 48 participants will be enrolled in the study. Participant follow-up will continue up to 3 years after the last participant is randomized. The estimated accrual period will be 12 months corresponding to an approximate total study duration of 4 years.

ELIGIBILITY:
Inclusion Criteria:

1. Participant must be ≥18 years or older.
2. Documented diagnosis of Multiple Myeloma (MM) as per International Myeloma Working Group (IMWG) criteria.
3. Must have at least ONE aspect of measurable disease, defined as one of the following:

   1. Urine M-protein excretion ≥200 mg/24 hrs (≥0.2 g/24 hrs), or
   2. Serum M-protein concentration ≥0.5 g/dL (≥5.0 g/L), or
   3. Serum Free Light Chain (FLC) assay: involved FLC level ≥10 mg/dL (≥100 mg/L) and an abnormal serum FLC ratio (<0.26 or >1.65).
4. Eastern Cooperative Oncology Group performance status of 0-2.
5. Adequate organ system function as defined by the below laboratory assessments. Hematologic

   1. Absolute neutrophil count (ANC) ≥1.5 X 109/L; granulocyte colony stimulating factor use within the past 14 days is NOT permitted.
   2. Hemoglobin ≥8.0 g/dL; transfusions within the past 14 days are NOT permitted. Erythropoietin use is allowed.
   3. Platelet count ≥50 x 109/L if Bone Marrow (BM) is >50% involved in myeloma. Otherwise ≥75 x 109/L; transfusions within the past 14 days are NOT allowed to reach this level.

   Hepatic
   1. Total bilirubin ≤1.5xULN (isolated bilirubin ≥1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
   2. Alanine aminotransferase (ALT) ≤ 2.5xUpper Limit of Normal (ULN). Renal

   <!-- -->

   1. Estimate glomerular filtration rate (eGFR) ≥30 mL/min/1.73 m2; calculated using the Modified Diet in Renal Disease (MDRD) formula.
   2. Spot urine (albumin/creatinine ratio) ≤500 mg/g (56 mg/mmol) OR
   3. Urine Dipstick: Negative trace; if ≥1+ only eligible if confirmed ≤500 mg/g [56 mg/mmol] by albumin/creatinine ratio (spot urine from first void).
6. Female participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies:

   A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:
   * Is not a woman of childbearing potential (WOCBP) defined as follows:

     1. ≥45 years of age and has not had menses for > 1 year
     2. Participants who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
     3. Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure.

        OR
   * Is a WOCBP and using two methods of reliable birth control (one method that is highly effective and one additional effective [barrier] method), beginning 4 weeks before initiating treatment with pomalidomide, during therapy, during dose interruptions, and continuing for 4 weeks following discontinuation of pomalidomide treatment. WOCBP participants must use one method of reliable birth control that is highly effective for 4 months following discontinuation of belantamab mafodotin or 3 months following the discontinuation of daratumumab. WOCBP must also agree not to donate eggs (ova, oocytes) for the purpose of reproduction during treatment, during dose interruptions and for 28-days following the last dose of pomalidomide or 3 months following discontinuation of daratumumab treatment or 4 months following discontinuation of belantamab mafodotin treatment whichever is longer.

   A WOCBP must have two negative pregnancy tests before therapy initiation. The first test should be performed within 10-14 days and the second test within 24 hours before the start of pomalidomide therapy.

   The participant should not receive pomalidomide until the Investigator has verified that the results of these pregnancy tests are negative. The Investigator should evaluate the effectiveness of the contraceptive method in relationship to the first dose of study treatment. The Investigator is responsible for a review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a woman with a nearly undetected pregnancy.
7. Male participants: contraceptive use should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies:

   Male participants are eligible to participate if they agree to the following during the intervention period and until 28 days after the last dose of pomalidomide or 3 months following the discontinuation of daratumumab or 6 months after the last dose of belantamab mafodotin, whichever is longer, to allow for clearance of any altered sperm.

   • Refrain from donating sperm

   PLUS either:
   * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent, OR
   * Must agree to use contraception/barrier as detailed below:

   Agree to use a male condom, even if they have undergone a successful vasectomy, and female partner to use an additional highly effective contraceptive method with a failure rate of <1% per year as when having sexual intercourse with a woman of childbearing potential (including pregnant females).
8. Participants must be able to understand the study procedures and agree to participate in the study by providing written informed consent.
9. Participant must have received only 1 prior line of therapy (including lenalidomide) and be lenalidomide refractory at any lenalidomide dose (i.e., nonresponsive while on lenalidomide therapy, or progresses within 60 days of last therapy with lenalidomide).

Exclusion Criteria:

1. Peripheral neuropathy or neuropathic pain Grade 2 or higher, as defined by the National Cancer Institute, Common Toxicity Criteria for Adverse Events (NCI CTCAE) Version 5.
2. Major surgery within 4 weeks before the first dose of study drug

   * NOTE 1: participant must be clinically stable following a major surgery to be entered in the study.
   * NOTE 2: major surgery shall be defined based on the Investigator's judgment according to the extent and complexity of the procedure, its pathophysiological consequences and consecutive clinical outcomes.
3. Presence of active renal condition (infection, requirement for dialysis, or any other significant condition that could affect participant's safety). Participants with isolated proteinuria resulting from MM are eligible, provided that they fulfil the other inclusion criteria.
4. Any serious and/or unstable pre-existing medical or psychiatric disorder, or other conditions (including laboratory abnormalities) that could interfere with participant's safety, obtaining informed consent, or compliance to the study procedures.
5. Evidence of active mucosal or internal bleeding uncontrolled by local therapy and not explained by reversible coagulopathy.
6. Current active unstable liver or biliary disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices, persistent jaundice, or cirrhosis (except for Gilbert's syndrome or asymptomatic gallstones; otherwise, stable non-cirrhotic chronic liver disease; or hepatobiliary involvement of malignancy as per the Investigator's assessment).
7. Participants with previous or concurrent malignancies other than MM are excluded. Exceptions are surgically treated cervical carcinoma in situ, or any other malignancy that has been considered medically stable for at least 2 years. The participant must not be receiving active therapy, other than hormonal therapy for this disease.

   * NOTE: Participants with curatively treated non-melanoma skin cancer are allowed without a 2-year restriction.
8. Evidence of cardiovascular risk including any of the following:

   * Evidence of current clinically significant untreated arrhythmias, including clinically significant electrocardiogram (ECG) abnormalities, second degree (Mobitz Type II), or third degree atrioventricular block.
   * Screening 12-lead ECG showing a baseline QT interval >470 msec
   * History of myocardial infarction, acute coronary syndromes (including unstable angina), coronary angioplasty, or stenting or bypass grafting within 3 months of Screening.
   * Class III or IV heart failure as defined by the New York Heart Association functional classification system
   * Uncontrolled hypertension.
9. Participant has known chronic obstructive pulmonary disease (COPD) (defined as a forced expiratory volume in 1 second [FEV1] <50% of predicted normal), persistent asthma, or a history of asthma within the last 2 years (controlled intermittent asthma or controlled mild persistent asthma is allowed).

   NOTE: Participants with known or suspected COPD must have a FEV1 test at screening.
10. Active infection requiring treatment.
11. Known human immunodeficiency virus infection, unless the participant can meet all of the following criteria:

    * Established anti-retroviral therapy for at least 4 weeks and HIV viral load <400 copies/mL.
    * CD4+ T-cell (CD4+) count ≥350 cells/uL.
    * No history of AIDS-defining opportunistic infections within the last 12 months.

      * NOTE: consideration must be given to ART and prophylactic antimicrobials that may have a drug:drug interaction and/or overlapping toxicities with belantamab mafodotin or other combination products as relevant
12. To be seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]) at screening or within 3 months prior to first dose of study treatment.

    * NOTE 1: Participants with resolved infection (i.e., participants who are positive for antibodies to hepatitis B core antigen [antiHBc] or antibodies to hepatitis B surface antigen [antiHBs]) must be screened using real-time polymerase chain reaction (PCR). Those who are PCR positive will be excluded.
    * NOTE 2: presence of antiHBs indicating previous vaccination will not constitute an exclusion criterion.
13. Positive hepatitis C antibody test result or positive hepatitis C RNA test result at screening or within 3 months before the first dose of study treatment unless the participant can meet the following criteria:

    * RNA test negative
    * Successful anti-viral treatment (usually 8 weeks duration) is required, followed by a negative hepatitis C virus (HCV) RNA test after a washout period of at least 4 weeks.
14. Current corneal epithelial disease except for mild punctate keratopathy.

    * NOTE: Participants with mild punctate keratopathy are allowed.
15. Intolerance or contraindications to anti-viral prophylaxis.
16. Unable to tolerate antithrombotic prophylaxis.
17. Active or history of venous thromboembolism within past 3 months.
18. AL amyloidosis (light chain amyloidosis), active POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal plasma proliferative disorder, skin changes) or active plasma cell leukemia at the time of screening.
19. Exhibiting clinical signs of or with a known history of meningeal or central nervous system involvement by MM.
20. Known intolerance or immediate or delayed hypersensitivity reaction or idiosyncratic reaction to: drugs chemically related to belantamab mafodotin, or any of the components of the study treatment; daratumumab subcutaneous (SC) or to any of its excipients; or infused protein products, sucrose, histidine, and polysorbate 80.
21. Use of an investigational drug within 14 days or 5 half-lives (whichever is longer) preceding the first dose of study drug.
22. Participant who has received prior treatment with daratumumab, pomalidomide or belantamab mafodotin will be excluded.

    * NOTE: Participants who received induction treatment with daratumumab (max 4 cycles) will be allowed as long as 6 months have passed since their treatment with daratumumab and cycle 1 day 1 (C1D1).
23. Plasmapheresis within 7 days before the first dose of study drug.
24. Participants with uncontrolled skin disease.
25. Participant must not have received a live or live-attenuated vaccine within 30 days prior to first dose of belantamab mafodotin.
26. Participant should not use contact lenses while receiving belantamab mafodotin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-10-20 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Part 1: Dose-Limiting Toxicity (DLT) | Up to 28 days
  The number (percent) of participants with DLTs using the DLT evaluable population.
Part 1 and 2: Adverse Events (AEs) and Serious adverse events (SAEs) | Up to 4 years
  The number (percent) of participants with AEs and SAEs using the DLT evaluable and Safety populations.
Part 1 and 2: Ocular Toxicity | Up to 4 years
  The number (percent) of participants with Grade ≥2 ocular toxicity per Keratopathy Visual Acuity (KVA) scale.
Part 2: Overall Response Rate (ORR) | Up to 4 years
  ORR as per IMWG by Investigator assessment; defined as the percentage of participants with a confirmed partial response (PR), very good partial response (VGPR), complete response (CR) or stringent CR (sCR) (For the 'intention to treat' (ITT) population).

SECONDARY OUTCOMES:
Part 1 and 2: Cumulative dose of belantamab mafodotin | Up to 4 years
  Cumulative belantamab mafodotin dose of (DLT evaluable population, safety population) administered in combination with daratumumab, pomalidomide and dexamethasone, i.e., the total dose of belantamab mafodotin that was administered.
Part 1: Overall Response Rate (ORR) | Up to 4 years
  ORR and 95% CI as per IMWG by Investigator Assessment (ITT population); ORR is defined as the percentage of participants with a confirmed PR, VGPR, CR or sCR.
Part 1: Very good partial response (VGPR) | Up to 4 years
  VGPR+ and 95% CI as per IMWG by Investigator Assessment (ITT population);ORR is defined as the percentage of participants with a confirmed VGPR, CR or sCR.
Part 1 and 2: Time to response (TTR) | Up to 4 years
  TTR as per IMWG by Investigator Assessment (ITT population). TTR is defined as the time (in months) between the date of randomization and the first evidence of confirmed response (PR or better) for participants who achieve a response (i.e., confirmed PR or better).
Part 1 and 2: Duration of Response | Up to 4 years
  DoR as per IMWG by Investigator Assessment (ITT population). DoR is defined as the time (months) from first evidence of confirmed PR or better until the earliest date of: documented disease progression (PD) per IMWG response criteria; or death due to PD among participants who achieved a response of PR or better. For alive and progression-free participants, data will be censored at the date of initiation of the subsequent line of treatment or at the last date of follow-up that the participant was known to be alive and progression-free.
Part 1 and 2: Complete Response Rate (CRR) | Up to 4 years
  CRR as per IMWG by Investigator Assessment (ITT population). CRR is defined as the percentage of participants with a confirmed CR or sCR. The denominator will be the total number of participants in each population and group respectively.
Part 1 and 2: Minimal Residual Disease (MRD) negative rate | Up to 4 years
  MRD negativity rate (ITT population); defined as the number (percent) of participants who achieve MRD negativity (at or below the threshold of 10-5), assessed via NGF in participants with CR or better response. The denominator will be the total number of participants in each population group respectively.
Part 1 and 2: Very Good Partial Response (VGPR) or better | Up to 4 years
  VGPR or better as per IMWG by Investigator Assessment (ITT population). VGPR or better rate is defined as the percentage of participants with a confirmed VGPR, CR or sCR. The denominator will be the total number of participants in each population, and group respectively.
Part 1 and 2: Progression Free Survival (PFS) | Up to 4 years
  PFS as per IMWG by Investigator Assessment (ITT population, Safety population). PFS is defined as the time (in months) from randomization until the earliest date of documented PD per IMWG, or death due to any cause. For participants who neither progress nor die, the PFS will be censored at the date of their last adequate disease assessment. For participants who start a new anti-myeloma treatment, PFS will be censored at the date of the last adequate assessment before the start of the new treatment. For a randomized participant who does not have any post-baseline disease assessments and who has not died, PFS will be censored at the randomization date.
Part 1 and 2: Overall Survival (OS) | Up to 4 years
  OS (ITT population, Safety population). OS is defined as the time from first dose/randomization until death due to any cause. If a participant is not known to have died, survival time will be censored at the date of last contact ("last known date alive").
Part 1 and 2: Abnormal ocular findings | Up to 4 years
  Number (percent) of participants with abnormal ocular findings (on ophthalmic exam) (DLT evaluable population, Safety population).
Part 1 and 2: Pharmacokinetics Analysis (PK population) | Up to 4 years
  Concentration-time data: linear and semi-logistic unique profiles of concentration-time and the mean and median profiles (as applicable) will be graphically represented for belantamab mafodotin. Belantamab mafodotin concentrations will be presented for each participant and summarized (as applicable) at each PK timepoint.
Part 2: Number of Ocular Symptoms and Related Impact | Up to 4 years
  Number of participants with within-participant meaningful change in ocular symptoms and related impacts as measured by the Vision Related Anamnestic Tool.
Part 2: Proportion of Ocular Symptoms and Related Impact | Up to 4 years
  Proportion of participants with within-participant meaningful change in ocular symptoms and related impacts as measured by the Vision Related Anamnestic Tool.
Part 1 and 2: Frequency of KVA Events | Up to 4 years
  No statistical comparison will be made between the 2 groups.
Part 1 and 2: Proportion of KVA Events | Up to 4 years
  No statistical comparison will be made between the 2 groups.
Part 1 and 2: Frequency of Dose holds | Up to 4 years
  No statistical comparison will be made between the 2 groups.
Part 1 and 2: Proportion of Dose holds | Up to 4 years
  No statistical comparison will be made between the 2 groups.
Part 1 and 2: Frequency of Worst Post-Baseline BCVA | Up to 4 years
  No statistical comparison will be made between the 2 groups.
Part 1 and 2: Proportion of Worst Post-Baseline BCVA | Up to 4 years
  No statistical comparison will be made between the 2 groups.
Part 1 and 2: Frequency of Grade 4 corneal findings | Up to 4 years
  No statistical comparison will be made between the 2 groups.
Part 1 and 2: Proportion of Grade 4 corneal findings | Up to 4 years
  No statistical comparison will be made between the 2 groups.

CONTACTS AND LOCATIONS:
Overall Officials: Evangelos Terpos, Prof, Principal Investigator — Department of Clinical Therapeutics, School of Medicine, National Kapodistrian University of Athens (NKUA)

IPD SHARING:
Plan to Share IPD: No